CLINICAL TRIAL: NCT00230321
Title: A Study of Darbepoetin Alfa in Patients With Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter L Greenberg (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Peter L Greenberg, Professor Emeritus, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEMMDS0001; HEMMDS0001; NCT00230321; 13536 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Blood Cancer; Myelodysplastic Syndromes; Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes | interventions — Darbepoetin alfa

ARMS (1):
- Darbepoetin alfa (Experimental): During the induction phase, the investigational agent DARBEPOETIN ALFA will be initiated at a dose of 4.5 ug/kg/week subcutaneously for 6 weeks. The dosage for the remaining treatment is dependent of patients response during the induction phase.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — During the induction phase, the investigational agent DARBEPOETIN ALFA will be initiated at a dose of 4.5 ug/kg/week subcutaneously.If patients do not achieve a major erythroid response by 6 weeks, the dose of DARBEPOETIN ALFA will be doubled to 9.0 ug/kg/week.

SUMMARY:
The primary objectives of the trial are to assess erythroid response to darbepoetin alfa, as determined by changes in hemoglobin and/or red blood cell (RBC) transfusion-dependence and to describe the safety profile of darbepoetin alfa in patients with MDS. The secondary objective is to assess bone marrow progenitor BFU-E growth before and after treatment with darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:- Diagnosis:

* Bone marrow aspirate/biopsy-proven MDS for > 2 months prior to enrollment.
* MDS French-American-British (FAB) subtypes refractory anemia (RA), RA with ringed sideroblasts (RARS), RA with excess blasts (RAEB), and non-proliferative chronic myelomonocytic leukemia (CMML) [WBC < 12,000/ml].
* Patients must have an untransfused hemoglobin < 10.0 g/dL and/or patients must be red cell transfusion-dependent for a period of at least 2 months prior to study entry.

  - Laboratory:
* Bilirubin < or = to 2 mg/dL
* ALT/SGPT < or = to 2.5 x the upper limit of normal (ULN)
* Normal renal function (Stanford: serum creatinine < 1.2 mg/dL [male], < 1.0 mg/dL [female]; Vanderbilt: < 1.5 mg/dL).

  * Age: > or = to 18
  * Other:
* ECOG performance status 0-2.
* Patients may receive standard supportive care, including transfusions and antibiotics as required.
* Patients must be r-HuEPO naive or must not have received prior treatment with r-HuEPO > or = to 40,000 U/week for more than 4 weeks. Exclusion Criteria:- Patients with secondary MDS or prior allogeneic bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2002-02; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
hemoglobin and/or red blood cell (RBC) transfusion-dependence.
To assess erythroid responses to DARBEPOETIN ALFA, as determined by changes in

SECONDARY OUTCOMES:
To assess bone marrow progenitor BFU-E growth before and after treatment
DARBEPOETIN ALFA

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Greenberg, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States